CLINICAL TRIAL: NCT05034978
Title: Point-of-care Testing for Improving the Detection of SARS-CoV-2 Infection in Healthcare Setting
Brief Title: Novel SARS-CoV-2 Point-of-care Testing
Status: Terminated | Type: Observational
Why Stopped: failure in enrolling eligible subjects during COVID-19 outbreaks
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shui-Shan Lee, MD, Research Professor, Chinese University of Hong Kong
Other Study IDs: Protocol HK POCT study
Record Dates: First submitted 2021-08-29; First posted 2021-09-05 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: SARS-CoV2 Infection
Keywords: SARS-CoV-2; point-of-care testing; rapid diagnostics; Hong Kong
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — evaluating the performance of a novel point-of-care test

SUMMARY:
The aim of the project is to study the feasibility of implementing a novel point-of-care test (POCT) for rapid detection of SARS-CoV-2 infection. A CRISPR-based detection kit would be piloted for testing of suspected SARS-CoV-2 infection in healthcare setting, with the objectives of evaluating the performance of the new test in the detection of SARS-CoV-2, and assessing the practicability of the new test for diagnosing SARS-CoV-2 infection in healthcare settings.

DETAILED DESCRIPTION:
A CRISPR-based lateral flow assay (LFA) detection kit would be designed and developed for testing for the presence of SARS-CoV-2. The aim of the project is to study the feasibility of implementing the novel point-of-care test (POCT) for rapid detection of SARS-CoV-2 infection in health service setting, with the following objectives: (b) Evaluation of the performance of novel POCT in comparison with conventional quantitative PCR in diagnosis SARS-CoV-2 infection and (c) Assessment of the practicability of LFA-CRISPR-based tests in the operating environments in healthcare settings.

Patients who are admitted to the isolation wards of Prince of Wales Hospital, Hong Kong would be invited to join the study. A total of 600 persons with suspected SARS-CoV-2 infection presenting with different symptomatology and epidemiological history will be recruited. Nasal, deep saliva and/or mouth gargle samples will be collected from all recruited subjects in accordance with standard clinical protocol. The samples would be tested for SARS-CoV-2 by the new Point-of-care test, in parallel with standard diagnostic testing of the hospital.

ELIGIBILITY:
Inclusion Criteria:

* adult patients admitted to isolation wards of the hospital who are
* of age of 18 or above;
* presentation with symptoms of COVID-19 and/or
* demonstration of exposure risk to SARS-CoV-2 infection.

Exclusion Criteria:

* inability to communicate in English or Chinese;
* known history of mental illness;
* prisoners.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: persons with exposure risk to SARS-CoV-2 infection who subsequently test positive or negative to conventional PCR-based testing for the diagnosis of the infection.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Test performance | 1 year
  agreement of point-of-care test result and conventional test

CONTACTS AND LOCATIONS:
Locations (1):
- Stanley Ho Centre for Emerging Infectious Diseases, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual participants data are not collected